CLINICAL TRIAL: NCT04292652
Title: Treatment With Endovascular or Open Repair for AAA - Comparison of Perioperative Myocardial Injury Detected With Holter-ECG and Troponin
Brief Title: Myocardial Injury in Treatment of AAA
Acronym: TREATROP
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Örebro University, Sweden (Other); Karlstad Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GoteborgU 01-20
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Aortic Aneurysm, Abdominal; Complication of Surgical Procedure; Myocardium; Ischemic
Keywords: AAA; Myocardial ischemic injury; Troponin; Holter-ECG; Vascular surgery
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EVAR group: Individuals undergoing endovascular aortic repair. n=40
  Interventions: Procedure: AAA surgery
- OR group: Individuals undergoing open repair. n=40
  Interventions: Procedure: AAA surgery

INTERVENTIONS:
Procedure: AAA surgery — EVAR is a mini invasive procedure to exclude aortic aneurysms with the intention to prevent rupture. Open repair is the traditional open surgical procedure for the same condition.

SUMMARY:
Comparison of elective infrarenal aneurysm surgery with open and endovascular technique, respectively, for subclinical ischemic myocardial injury detectable with troponin T and/or 3-channel Holter ECG with ST analysis

DETAILED DESCRIPTION:
Background: Traditional open surgery for abdominal aortic aneurysm (AAA) is burdened with complication risk from several organ systems, and also mortality figures of 3.5 - 5.5%. Over 50% of early mortality can be attributed to cardiovascular complications. Myocardial infarction is the dominant organ-specific cause of both early and late mortality in patients operated on for AAA. Endovascular surgery (EndoVascular Aortic Repair, EVAR) was developed during the 90's as an alternative method that is considered less invasive and more well-tolerated from a cardiovascular perspective.

Troponin T is a very sensitive and specific marker that predicts mortality in patients with acute symptoms of unstable angina and/or heart attack. Previous studies have also shown a high incidence of elevated troponin levels in patients who underwent major surgical procedures, especially vascular surgery, even in the absence of corresponding clinical or ECG-related symptoms of cardiac muscle injury. Several studies have also demonstrated that elevated troponin levels after surgery predict increased morbidity and mortality both short-term and long-term.

Objective: To prospectively compare elective open and endovascular surgery of AAA with respect to myocardial injury detectable with troponin T. Furthermore, to compare open and endovascular AAA surgery for the total number of periods of oxygen deficiency in cardiac muscle during and at early stages after surgery using a special ECG method (48-hour 3-channel Holter ECG with ST analysis).

Main aim of the study: To assess whether EVAR induce less myocardial injury compared with open repair for AAA.

Significance: Myocardial infarction is the predominant cause of mortality in open surgical procedure for AAA. In several previous studies, troponin T rise has been associated with impaired both short-term and long-term prognosis in elderly patients undergoing major elective surgery. This study may provide information on whether the endovascular technique provides a reduction in myocardial injury, measured as elevated troponin T or myocardial ischemia with 3-channel Holter ECG. In this way, our study can provide improved decision support in the choice of the most appropriate treatment method in the individual case.

ELIGIBILITY:
Inclusion Criteria:

* Accepted for AAA surgery of either one of the operative techniques

Exclusion Criteria:

* High anesthesiological risk
* Preoperative cardiac condition with EF < 25 or ischemic signs on preoperative evaluation
* Severe renal insufficiency with s-creatinine >200

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive individuals accepted for either open or endovascular aortic repair in two Swedish hospitals
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Ischemic myocardial injury | Perioperative
  Perioperative myocardial injury induced by the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Per Skoog, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Gothenburg university, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No